CLINICAL TRIAL: NCT03571711
Title: Single- and Multiple-dose Pharmacokinetics of Meropenem in Spontaneous Bacterial Peritonitis and Liver Cirrhosis
Brief Title: Meropenem Pharmacokinetics in Spontaneous Bacterial Peritonitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: SBP-MER-PK-2018
Record Dates: First submitted 2018-05-28; First posted 2018-06-27 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Peritonitis Bacterial; Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Meropenem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Plasma and ascites samples are taken before 30, 60, 120, 240, 480, 510, 540, 600, 720, 960, 990, 1020, 1080, 1200 and 1440 minutes after the first meropenem Infusion at day one and four after study enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Meropenem therapy in SBP: Patients in a tertiary care Hospital with meropenem injection due to spontaneous bacterial Peritonitis.
  Interventions: Drug: Meropenem Injection

INTERVENTIONS:
Drug: Meropenem Injection — Meropenem is administered as prescribed by treating physician

SUMMARY:
The emergence of multidrug-resistant bacteria has increased the use of meropenem in spontaneous bacterial peritonitis (SBP). Additionally, recent studies suggested female gender as an independent risk factor for mortality in SBP. Studies regarding possible sex dependent differences in meropenem pharmacokinetics in SBP are scarce. The aim of this study is to determine the pharmacokinetics of meropenem during SBP in female and male patients with liver cirrhosis to investigate whether pharmacodynamics therapy goals are met.

DETAILED DESCRIPTION:
Spontaneous bacterial Peritonitis (SBP) in liver cirrhosis is a severe and increasingly common disease, which is associated with high morbidity, mortality and high costs for the investigator's health care system. In addition to age and severity of comorbidities, female sex is associated with detrimental outcome. Delayed diagnosis and therapy of SBP may lead to a higher mortality in this patient population. Therefore, an early diagnosis and adequate anti-infective therapy is essential. Due to the accumulation of antimicrobial-resistant (AMR) pathogens, especially in nosocomial SBP, empirical application of broad-spectrum antibiotics is recommended in the therapy of SBP.During the use of antibiotic drugs in general, pharmacokinetic/pharmacodynamic (PK/PD) targets, as the achieved time period over the minimal inhibitory concentration (MIC), should be evaluated to increase drug efficacy and reduce AMR development. Pharmacokinetic studies of meropenem concentrations at the infection site in this particular group of patients are rare in the literature. Recent studies in critically ill patients showed highly variable meropenem concentrations in peritoneal fluid after iv administration. The aim of this study is to determine the pharmacokinetics of meropenem during SBP in female and male patients with liver cirrhosis to investigate whether pharmacodynamics therapy goals are met.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 years
* Administration of meropenem
* Diagnosis of liver cirrhosis
* Diagnosis of spontaneous bacterial Peritonitis
* Indication for peritoneal drainage catheter

Exclusion Criteria:

* Incapacity to give informed consent
* Participation in other studies
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in a tertiary care Hospital with meropenem therapy due to spontaneous bacterial Peritonitis.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2018-06-28 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Peak concentrations of meropenem in single- and multiple-dose pharmacokinetics | 5 days
  Single- and multiple-dose pharmacokinetic measurements of meropenem concentrations in blood plasma and ascites fluid and evaluation of Peak Levels concentrations in blood plasma and ascites fluid and evaluation of peak concentrations.
Area under the curve of meropenem in single- and multiple-dose pharmacokinetics | 5 days
  Single- and multiple-dose pharmacokinetic measurements of meropenem concentrations in blood plasma and ascites fluid and evaluation of area under the curve characteristics
Trough concentrations of meropenem in single- and multiple-dose pharmacokinetics | 5 days
  Single- and multiple-dose pharmacokinetic measurements of meropenem concentrations in blood plasma and ascites fluid and evaluation of trough concentrations.
Time over MIC of meropenem in single- and multiple-dose pharmacokinetics | 5 days
  Single- and multiple-dose pharmacokinetic measurements of meropenem concentrations in blood plasma and ascites fluid and evaluation of achieved time period with drug concentration above the minimal inhibitory concentration breakpoint of 8 mg/L.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Maasoumy, PD Dr., Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany